

## **CONSENT FORM**

| Full title of Project: Glycaemic Re | esponse (GR) and Ins | ulin Response (IR) | testing of foods |
|---|---|---|---|
|---|---|---|---|

Contacts:

Isabel Butler, Manager, Oxford Brookes Centre for Nutrition and Health (OxBCNH)

Dr. Sangeetha Thondre, Senior Lecturer and Research Lead

OxBCNH
Department of Sport, Health Sciences and Social Work
Faculty of Health and Life Sciences
Oxford Brookes University
Gipsy Lane Campus
Oxford OX3 0BP

Tel: 01865 483297 / 01865 483988

Email: <a href="mailto:ibutler@brookes.ac.uk">ibutler@brookes.ac.uk</a> / <a href="mailto:pthondre@brookes.ac.uk">pthondre@brookes.ac.uk</a> / <a href="mailto:pthondre@brookes.ac.uk">pthondre@brookes.ac.uk</a> / <a href="mailto:pthondre@brookes.ac.uk">pthondre@brookes.ac.uk</a> / <a href="mailto:pthondre@brookes.ac.uk">pthondre@brookes.ac.uk</a> <a href="mailto:pthondr

## Please initial box

| 1. | I confirm that I have read and understand the information sheet for the above study and have had the opportunity to ask questions. | | |
|---|---|---|---|
| 2. | I understand that my participation is voluntary and that I am free to withdraw at any time, without giving reason. | | |
| 3. | I agree to take part in the above s | study. | |
| —<br>Na | me of Participant | Date | Signature |
| Na | me of Researcher | Date | Signature |



## Receipt of signed consent form

| I confirm that I have received a signed copy of the consent form overleaf. | | |
|---|---|---|
| Name of Participant | Date | Signature |